CLINICAL TRIAL: NCT01172626
Title: Exploration of Genotype Based Personalized Prescription of Valproate Sodium in Anti-epileptic Treatment
Acronym: EGBPPVPA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: School of Pharmaceutical Sciences, Sun Yat-sen University ( Min Huang ), Sun Yat-sen University
Other Study IDs: VPA20100716
Record Dates: First submitted 2010-07-29; First posted 2010-07-30 (Estimated); Last update posted 2010-07-30 (Estimated); Status verified 2010-07

CONDITIONS: Epilepsy; Adverse Effects
Keywords: epilepsy; valproate sodium; metabolic enzymes; adverse effects; systemic adverse effects
MeSH Terms: conditions — Epilepsy | interventions — Valproic Acid; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood for DNA extraction as well as for pharmacokinetic studies
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- epileptic patients: epileptic patients receiving treatment with continuous Sodium Valproate
  Interventions: Drug: valproate sodium; Genetic: Polymorphism Analysis; Other: Pharmacokinetic analysis

INTERVENTIONS:
Drug: valproate sodium — oral administration,15-30mg/kg,daily
  Other Names: Depakine
Genetic: Polymorphism Analysis — Analysis of genetic polymorphisms of the drug metabolic enzymes involving in the deactivation and elimination of Valproate sodium
Other: Pharmacokinetic analysis — laboratory analysis of concentration of Valproate sodium and 4-ene-Valproate in plasma
  Other Names: concentration detection method

SUMMARY:
The purpose of this study is to investigate the relationship between the side effects of valproate sodium in the treatment of epilepsy in Han Chinese and the genetic polymorphisms of drug metabolizing enzymes and pharmacokinetics of valproate sodium.

DETAILED DESCRIPTION:
Valproate sodium is a widely applied agent in the treatment of epilepsy. Although Valproate sodium is effective in clinic, it is able to induce several side effects, including weight gain, thinned hair, loss of appetite, nausea, vomiting, hepatotoxicity, hematotoxicity, thrill, etc. However, the remarkable variability of the reactions to the drug -- the incidence of side effect or the outcome of the treatment -- has been observed among patients. Valproate sodium is metabolized by some enzymes in the liver to transform it into several unreactive chemicals for excretion. Among them there are two toxic metabolites catalyzed by the specific metabolic enzymes. This study is designed to explore the genetic variation among individuals in the key processes of the deactivation and elimination of Valproate sodium in order to find out whether these genetic factors are associated to the side effects or efficacy. The further understanding into the factors concerning on the drug might imply possible solution to minimize the incidence of side effects in epileptic patients.

ELIGIBILITY:
Inclusion Criteria:

* The patients must have been diagnosed as epilepsy according to The International League Against Epilepsy (ILAE) criteria published in 2001.
* The patients must sign the informed consent. And for the patients who are under 18 years old, both the signatures of their legal guardians and that of the patients are required on the written informed consent.
* The patients are receiving the regimen of 15-30mg/kg valproate sodium given as daily oral administration.

Exclusion Criteria:

* Pregnant women, women in breast-feeding period and the women who refuse to take contraception measures during treatment.
* Patients with poor compliance.
* Patients who have blood transfusion during the therapy.

Ages: 4 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients receiving treatment with valproate sodium
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2010-08; Primary Completion 2013-03 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
epileptic seizure | one year

CONTACTS AND LOCATIONS:
Overall Officials: Huang Min, PhD, Study Chair — Institute of Clinical Pharmacology, School of Pharmaceutical Sciences, Sun Yat-sen University, Guangzhou, China; Wang Xueding, PhD, Study Director — Institute of Clinical Pharmacology, School of Pharmaceutical Sciences, Sun Yat-sen University, Guangzhou, China; Chen Zhuojia, PhD, Principal Investigator — Institute of Clinical Pharmacology, School of Pharmaceutical Sciences, Sun Yat-sen University, Guangzhou, China; Zhou Jueqian, MMSC, Study Director — Department of Neurology, the First Affiliated Hospital, Sun Yat-sen University, Guangzhou, China; Fang Ziyan, MMSC, Principal Investigator — Department of Neurology, the First Affiliated Hospital, Sun Yat-sen University, Guangzhou, China
Locations (1):
- Institute of Clinical Pharmacology, School of Pharmaceutical Sciences, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Chen J, Su QB, Tao YQ, Qin JM, Zhou Y, Zhou S, Li HL, Chen ZJ, Zhou YF, Zhou LM, Wang XD, Huang M. ABCC2 rs2273697 is associated with valproic acid concentrations in patients with epilepsy on valproic acid monotherapy. Pharmazie. 2018 May 1;73(5):279-282. doi: 10.1691/ph.2018.7344. PMID 29724294